CLINICAL TRIAL: NCT02480920
Title: Drug Adherence in Patients Taking New Oral Anticoagulation Therapy in Turkey
Brief Title: Adherence to New Oral Anticoagulation Therapy in Turkey
Acronym: NOAC-TR
Status: Completed | Type: Observational
Sponsor: Cardiovascular Academy Society, Turkey (Other)
Responsible Party: Sponsor
Other Study IDs: NOAC-TR
Record Dates: First submitted 2015-06-19; First posted 2015-06-25 (Estimated); Results first posted 2019-01-31 (Actual); Last update posted 2019-04-09 (Actual); Status verified 2019-04

CONDITIONS: Atrial Fibrillation
Keywords: Atrial fibrillation Drug Adherence; New Oral Anticoagulants; Drug Adherence
MeSH Terms: conditions — Atrial Fibrillation; Medication Adherence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study will compose a national database of drug adherence and investigate the factors that affect drug adherence in patients taking new oral anticoagulation therapy in Turkish Population.

DETAILED DESCRIPTION:
NOACs have several clinical and pharmacological advantages over warfarin however suboptimal adherence is one of the most common causes of failure to respond to medications and outcomes.

This observational multicenter, retrospective study, will compose a national database of drug adherence and investigate the factors that affect drug adherence in patients taking new oral anticoagulation therapy in Turkey.

Social support and adherence to therapy factors that may affect drug adherence and adverse events will be assessed by self-report questionnaires.

Non-adherence will be tested for demographic, clinical, awareness of NOAC therapy and socioeconomic factors.

ELIGIBILITY:
Inclusion Criteria:

* Patients >18 years old
* Outpatients using a NOAC for at least 3 months duration, with a primary diagnosis of new-onset, non-valvular atrial fibrillation
* Patients signed patient informed sheet and informed consent form

Exclusion Criteria:

* Patients under 18 years old
* Patients refused to sign informed consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Outpatients using a NOAC for at least 3 months duration, with a primary diagnosis of new-onset, non-valvular atrial fibrillation
Sampling Method: Probability Sample
Enrollment: 2738 (Actual)
Dates: Start 2015-07; Primary Completion 2016-03 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Volkan Emren, MD, Principal Investigator — Cardiovascular Academy Society, İzmir, Turkey
Locations (1):
- Volkan Emren, Afyonkarahisar, Turkey (Türkiye)

RESULTS

PARTICIPANT FLOW:
Groups:
- Study Popülation: Who Received NOAC for More Than 3 Months: This multicenter cross-sectional study was conducted between September 2015 and February 2016 in 45 centers encompassing all the geographical regions of Turkey. A total of 3150 patients were evaluated in this study. The 163 patients with a sociocultural level inadequate to fill the questionnaire and the 249 patients who received new oral anticoagulant for less than 3 months were excluded from the study. This study was conducted with the remaining 2738 patients.
Period: Overall Study
Arm/Group | Study Popülation: Who Received NOAC for More Than 3 Months
Started | 2738
Completed | 2738
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Study Population: This multicenter cross-sectional study was consisted of patients who with non-valvular atrial fibrillation (NVAF) receiving Non-vitamin K antagonist oral anticoagulants NOACs), older than 18 years, who were followed up in cardiology clinics, and who received dabigatran (110-150 mg), rivaroxaban (15-20 mg), or apixaban (2.5-5 mg) for the last 3 months with >30 days of supply due to NVAF.
  The patients were categorized into 2 groups as adherent patients who had high and medium adherence (Morisky score 6 or more) and non-adherent patients who had low adherence (Morisky score 5 or less).
Arm/Group | Study Population
Number analyzed (Participants) | 2738
Age, Continuous [Mean (Standard Deviation); unit: years] | 70 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1623
  Male | 1115

OUTCOME MEASURES:

1. Primary Outcome: Compliance of NOACs in Turkish Population
Description: Factors that may affect drug adherence and adverse events will be assessed by self-report questionnaires. Non-adherence will be tested for demographic, clinical, awareness of NOAC therapy and socioeconomic factors.
  The validity of the Morisky Adherence Scale had already been demonstrated with regard to medication adherence in patients receiving vitamin K antagonists. An extended 8-item Morisky scale was used instead of the original 4-item Morisky scale in order to better identify the situations and the conditions that could affect medication adherence and to better assess the psychometric features.The reliability and the validity of the 8-item Morisky Adherence Scale translated into Turkish had been demonstrated in Turkish population by previous studies.
Time Frame: 10 months
Measure: Count of Participants; unit: Participants
Groups:
- Study Popülation: Who Received NOAC for More Than 3 Months: In order to identify the independent predictive variables that could affect the medication adherence of the patients with logistic regression analysis, the patients were categorized into 2 groups as adherent patients who had high and medium adherence (Morisky score 6 or more) and nonadherent patients who had low adherence (Morisky score 5 or less).
Arm/Group | Study Popülation: Who Received NOAC for More Than 3 Months
Number analyzed (Participants) | 2378
Participants
  low adherence | 1342
  high and medium adherence | 1036

ADVERSE EVENTS:
Groups:
- Advers Events: The adverse effects, stroke, and any bleeding complication during NOAC treatment. Major bleeding was defined as a hemorrhage leading to a reduction in hemoglobin concentration of 2 g/dL, necessitating the transfusion of 2 or more units of blood, or symptomatic bleeding into a critical area or organ.
Arm/Group | Advers Events
Serious Adverse Events (participants affected / at risk) | 687/2738
Other Adverse Events (participants affected / at risk) | 0/2738
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Advers Events (N=2738)
Stroke (Nervous system disorders) | 100
Bleeding (General disorders) | 577 — Any bleeding (major or minor) complication during NOAC treatment.
Systemic Embolism (Vascular disorders) | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No